CLINICAL TRIAL: NCT04202458
Title: Boosting REcanalization of Thrombectomy for Ischemic Stroke by Intra-arterial TNK (BRETIS-TNK): a Prospective, Random, Pilot Study
Brief Title: Boosting REcanalization of Thrombectomy for Ischemic Stroke by Intra-arterial TNK (BRETIS-TNK)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Professor, General Hospital of Shenyang Military Region
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: k(2019)29
Record Dates: First submitted 2019-12-15; First posted 2019-12-17 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intra-arterial tenecteplase administration (Experimental): Intra-arterial administration of 4mg tenecteplase is given after microcatheter navigation through the clot. Intra-arterial administration of tenecteplase (0.4 mg/min) continuously is given after the first attempt of thrombectomy device pass for 30 minutes, and then followed by DSA
  Interventions: Drug: intra-arterial tenecteplase administration

INTERVENTIONS:
Drug: intra-arterial tenecteplase administration — Intra-arterial administration of 4mg tenecteplase is given after microcatheter navigation through the clot. Intra-arterial administration of tenecteplase (0.4 mg/min) continuously is given after the first attempt of thrombectomy device pass for 30 minutes, and then followed by DSA.

SUMMARY:
Thrombolysis and endovascular thrombectomy are the most efficient treatments for acute ischemic stroke patients in time window. However, sufficient recanalization (mTICI2b-3) can 't be acquired in all patients under thrombectomy. The EXTEND-IA TNK study indicated that tenecteplase before thrombectomy was associated with a higher incidence of reperfusion and better functional outcome than alteplase among patients with ischemic stroke treated within 4.5 hours after symptom onset. This study intends to explore whether a combination of thrombectomy and intra-arterial TNK administration can increase recanalization rate after the first attempt of thrombectomy device pass for ischemic Stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Patients who presented with acute ischemic stroke and a large vessel occlusion in the anterior circulation and met the criteria of mechanical thrombectomy;
3. The subtype of ischemic stroke is large-artery atherosclerosis according to TOAST classification;
4. The availability of informed consent.

Exclusion Criteria:

1. Other sub-types of ischemic stroke such as cardioembolism.
2. Hemorrhagic stroke such as cerebral hemorrhage, subarachnoid hemorrhage.
3. Coagulation disorders, systematic hemorrhagic tendency, thrombocytopenia (<100000/mm3).
4. Severe hepatic or renal dysfunction, increase in ALT or AST (more than 2 times of upper limit of normal value), increase in serum creatinine (more than 1.5 times of upper limit of normal value) or requiring dialysis.
5. Severe uncontrolled hypertension (systolic blood pressure over 200mmHg or diastolic blood pressure over 110 mmHg).
6. Patients allergic to any ingredient of drugs in our study.
7. Unsuitable for this clinical studies assessed by researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Proportion of sufficient recanalization | Immediately after TNK treatment
  sufficient recanalization is defined as TICI 2b-3

SECONDARY OUTCOMES:
Proportion of favorable outcome | 90 days
  favorable outcome is defined as mRS 0-2
proportion of early neurological improvement | 48 hours
  early neurological improvement is defined as more than 4 decrease in NIHSS

OTHER OUTCOMES:
incidence of symptomatic intracranial haemorrhage | 48 hours
  more than 4 increase in NIHSS caused by intracranial bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao ZA, Qiu J, Wang L, Zhao YG, Sun XH, Li W, Liu X, Li XL, Liu L, Chen MR, Chen HS. Intra-arterial tenecteplase is safe and may improve the first-pass recanalization for acute ischemic stroke with large-artery atherosclerosis: the BRETIS-TNK trial. Front Neurol. 2023 Apr 18;14:1155269. doi: 10.3389/fneur.2023.1155269. eCollection 2023. PMID 37143999